CLINICAL TRIAL: NCT06268912
Title: Cryoanalgesia: Temperature Modulation for Pain Management in Irreversible Pulpitis a Randomized Clinical Trial
Brief Title: Cryoanalgesia for Irreversible Pulpitis
Acronym: CryPain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Gonzalo Gómez Val, Clinical Professor, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: END-ECL-2022-01; END-ECL-2022-01 (Other: UIC)
Record Dates: First submitted 2024-01-09; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pulpitis - Irreversible
Keywords: Cryoanalgesia; Irreversible Pulpitis; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cold Mepivacaine (Experimental): Mepivacaine 3% at 5ºC
  Interventions: Procedure: Cold Mepivacaine
- Mepivacaine at room temperature (Active Comparator): Mepivacaine 3% at room temperature
  Interventions: Procedure: Mepivacaine at room temperature

INTERVENTIONS:
Procedure: Cold Mepivacaine — change the temperature, 3% at 5ºC
  Arms: Cold Mepivacaine
Procedure: Mepivacaine at room temperature — no change the temperature of anesthesia
  Arms: Mepivacaine at room temperature

SUMMARY:
The aim of the present study was to evaluate the effectiveness of pulpal anesthesia in pain control during endodontic treatment by lowering the temperature of the injected plain 3% cold Mepivacaine (5ºC) compared to 3% Mepivacaine at room temperature in teeth with irreversible pulpitis.

DETAILED DESCRIPTION:
Mepivacaine has some advantages over other anesthetics. The investigators wanted to compare whether changing temperature could improve its effectiveness in cases of irreversible pulpitis.

ELIGIBILITY:
Inclusion Criteria:

All Patients within the age group of 18-100 years old,

* Patients diagnosed of irreversible pulpitis.

Exclusion Criteria:

* Moderate to pulp necrosis,
* Previous initiated treatment.
* Pregnancy or lactation.
* Allergy or problems to any substances used in the study,
* Acute apical abscess.
* Chronic apical abscess.
* Unrestorable teeth.
* Unsuccessful anesthesia technique (no lip numbness for lower molars or positive response to cold test).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2024-01-07 (Actual)

PRIMARY OUTCOMES:
Assessment of Pain and Anxiety | 1 visit of 1 hour
  Pain during injection, caries removal, access cavity, and instrumentation were recorded. The patients received a full description of the procedure, and patients were asked to rate their current pain and their anxiety with a descriptive scale (Heft-Parker Visual Analog Scale (VAS) before starting the treatment. A visual analog scale of 170 mm that the start points on the left side means "no pain" and the endpoint on the right side means "severe pain". The participants indicated their pain level by marking a point on the scale that best represented their experience. For data interpretation, the Visual Analog Scale (VAS) was segmented into four categories: no pain corresponded to 0 mm on the scale, mild pain as greater than 0 and ≤54mm, moderate pain defined as greater than 54 mm and less than 114 mm and severe pain defined as 114 mm or more.

CONTACTS AND LOCATIONS:
Overall Officials: gonzalo gomez, Principal Investigator — UIC
Locations (1):
- Gonzalo Gomez, Barcelona, Spain